CLINICAL TRIAL: NCT07109206
Title: Cardio-circulatory and Respiratory Monitoring for Prediction of Outcome in Mechanically Ventilated Chronic Obstructive Pulmonary Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Karim Osama Mohammed Sleem, Dr, Assiut University
Other Study IDs: KarimPhD1
Record Dates: First submitted 2025-06-23; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease); Cardiometry; Weaning Invasive Mechanical Ventilation
Keywords: Intensive-care, COPD, ICON, Weaning
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Success: Cases with successful weaning and extubation from mechanical ventilation
- Failed: Group with failed weaning trial

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) remains a leading cause of morbidity and mortality worldwide, often necessitating invasive mechanical ventilation (MV) during acute exacerbations. Weaning these patients from MV is a critical juncture in their care, as prolonged ventilation is associated with increased complications, including ventilator-associated pneumonia, diaphragmatic dysfunction, and higher healthcare costs. Traditional weaning indices, such as the Rapid Shallow Breathing Index (RSBI), Maximum Inspiratory Pressure (MIP), and the Integrative Weaning Index (IWI), New Integrative Weaning Index (NIWI) have been employed to predict weaning outcomes. However, their predictive accuracy in COPD patients is variable, often due to the heterogeneous nature of the disease and the presence of comorbidities. Recent advancements have introduced non-invasive hemodynamic monitoring tools, such as the ICON® (Electrical Cardiometry), which measures parameters like cardiac output, stroke volume, and thoracic fluid content. These parameters may offer additional insights into a patient's readiness for weaning by providing real-time data on cardiovascular and fluid status, which are crucial in the weaning process. There is a scarcity of data comparing the predictive value of ICON parameters with traditional weaning indices in COPD patients. Understanding whether ICON-derived metrics can enhance weaning predictions and lead to more individualized and effective weaning strategies, reducing the duration of MV and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All COPD patients who are mechanically ventilated for more than 48 h due to acute exacerbation and fulfilling weaning criteria will be included in the study.

Exclusion Criteria:

1. Patients younger than 18 years old.
2. Patients with pneumothorax, pleural, or pericardial effusion.
3. Patients with injuries, burns, or wounds which precludes the proper application of the device electrodes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: location: Assiut University Hospital Respiratory Intensive Care unit Population: All COPD patients admitted to Assiut University Hospital Respiratory Intensive Care unit, willingly sign informed consent, match the inclusion criteria and don't have a feature listed in the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate the accuracy of non-invasive hemodynamic parameters using Electric Cardiometry to predict weaning outcome in mechanically ventilated COPD patients. | 2 Years
  Assess the accuracy of the non-invasive hemodynamic parameters (Cardiac index, Thoracic fluid content, contractility, contractility index, systemic vascular resistance) using Electric Cardiometry device ICON® to predict the outcome of the weaning trial in mechanically ventilated COPD patients.

SECONDARY OUTCOMES:
Evaluate respiratory indices (RSBI, IWI, MIWI) as predictors of weaning outcome in mechanically ventilated COPD patients | 2 years
  Assess the accuracy of currently used respiratory indices (RSBI, IWI, MIWI) in the prediction of the outcome of weaning trial. These indices are currently used widely to predict the success or failure of weaning; However, there as still no consensus on a universal parameter and cut-off point.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Sleem, Master's Degree, Principal Investigator — Assiut University Medical School
Locations (1):
- Assiut University Medical School., Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hajian-Tilaki K. Receiver Operating Characteristic (ROC) Curve Analysis for Medical Diagnostic Test Evaluation. Caspian J Intern Med. 2013 Spring;4(2):627-35. PMID 24009950
- [Background] McHugh ML. The chi-square test of independence. Biochem Med (Zagreb). 2013;23(2):143-9. doi: 10.11613/bm.2013.018. PMID 23894860
- [Background] Paulus WJ. H2FPEF Score: At Last, a Properly Validated Diagnostic Algorithm for Heart Failure With Preserved Ejection Fraction. Circulation. 2018 Aug 28;138(9):871-873. doi: 10.1161/CIRCULATIONAHA.118.035711. No abstract available. PMID 30354456
- [Background] Pfeffer MA, Shah AM, Borlaug BA. Heart Failure With Preserved Ejection Fraction In Perspective. Circ Res. 2019 May 24;124(11):1598-1617. doi: 10.1161/CIRCRESAHA.119.313572. PMID 31120821
- [Background] Papadimitriou L, Georgiopoulou VV, Kort S, Butler J, Kalogeropoulos AP. Echocardiography in Acute Heart Failure: Current Perspectives. J Card Fail. 2016 Jan;22(1):82-94. doi: 10.1016/j.cardfail.2015.08.001. Epub 2015 Aug 13. PMID 26277267
- [Background] Fathy S, Hasanin AM, Raafat M, Mostafa MMA, Fetouh AM, Elsayed M, Badr EM, Kamal HM, Fouad AZ. Thoracic fluid content: a novel parameter for predicting failed weaning from mechanical ventilation. J Intensive Care. 2020 Mar 5;8:20. doi: 10.1186/s40560-020-00439-2. eCollection 2020. PMID 32161651
- [Background] Vahedian-Azimi A, Gohari-Moghadam K, Rahimi-Bashar F, Samim A, Khoshfetrat M, Mohammadi SM, de Souza LC, Mahmoodpoor A. New integrated weaning indices from mechanical ventilation: A derivation-validation observational multicenter study. Front Med (Lausanne). 2022 Jul 22;9:830974. doi: 10.3389/fmed.2022.830974. eCollection 2022. PMID 35935785
- [Background] Schmidt GA, Girard TD, Kress JP, Morris PE, Ouellette DR, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, Hough CL, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Truwit JD. Liberation From Mechanical Ventilation in Critically Ill Adults: Executive Summary of an Official American College of Chest Physicians/American Thoracic Society Clinical Practice Guideline. Chest. 2017 Jan;151(1):160-165. doi: 10.1016/j.chest.2016.10.037. Epub 2016 Nov 3. PMID 27818329
- [Background] Sungono V, Hariyanto H, Soesilo TEB, Adisasmita AC, Syarif S, Lukito AA, Widysanto A, Puspitasari V, Tampubolon OE, Sutrisna B, Sudaryo MK. Cohort study of the APACHE II score and mortality for different types of intensive care unit patients. Postgrad Med J. 2022 Dec 1;98(1166):914-918. doi: 10.1136/postgradmedj-2021-140376. PMID 37063012
- [Background] Abdelgawad TA, Ibrahim HM, Elsayed EM, Abdelhamid NS, Bawady SAH, Rezk AR. Hemodynamic monitoring during weaning from mechanical ventilation in critically ill pediatric patients: a prospective observational study. BMC Pediatr. 2024 Oct 26;24(1):681. doi: 10.1186/s12887-024-05110-5. PMID 39462317
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Zakarias D, Marics G, Kovacs K, Jermendy A, Vatai B, Schuster G, Toth-Heyn P, Szabo J A, Lodi C. [Clinical application of the electric cardiometry based non-invasive ICON(R) hemodynamic monitor]. Orv Hetil. 2018 Nov;159(44):1775-1781. doi: 10.1556/650.2018.31225. Hungarian. PMID 30392409
- [Background] Greiwe G, Saad R, Hapfelmeier A, Neumann N, Tariparast P, Saugel B, Flick M. Electrical cardiometry for non-invasive cardiac output monitoring: a method comparison study in patients after coronary artery bypass graft surgery. J Clin Monit Comput. 2025 Apr;39(2):371-376. doi: 10.1007/s10877-024-01246-y. Epub 2024 Dec 11. PMID 39661264
- [Background] Nemer SN, Barbas CS, Caldeira JB, Carias TC, Santos RG, Almeida LC, Azeredo LM, Noe RA, Guimaraes BS, Souza PC. A new integrative weaning index of discontinuation from mechanical ventilation. Crit Care. 2009;13(5):R152. doi: 10.1186/cc8051. Epub 2009 Sep 22. PMID 19772625
- [Background] Agusti A, Vogelmeier C, Faner R. COPD 2020: changes and challenges. Am J Physiol Lung Cell Mol Physiol. 2020 Nov 1;319(5):L879-L883. doi: 10.1152/ajplung.00429.2020. Epub 2020 Sep 23. No abstract available. PMID 32964724
- [Background] Huo Y, Guo S, Zhang K, Zhang T, Li B, Zhang Q, Han Y, Wang X, Hu Z. A clinical study on the ability of the integrative weaning index to predict weaning from mechanical ventilation. Ann Palliat Med. 2020 Sep;9(5):3162-3169. doi: 10.21037/apm-20-1335. PMID 33065782
- [Background] Gadre SK, Duggal A, Mireles-Cabodevila E, Krishnan S, Wang XF, Zell K, Guzman J. Acute respiratory failure requiring mechanical ventilation in severe chronic obstructive pulmonary disease (COPD). Medicine (Baltimore). 2018 Apr;97(17):e0487. doi: 10.1097/MD.0000000000010487. PMID 29703009